CLINICAL TRIAL: NCT03088852
Title: Magnesium Deficiency In Patients Hospitalized in Internal Medicine Wards
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Frieda Wolf (Other)
Responsible Party: Sponsor-Investigator, Frieda Wolf, Senior Physician in Internal Medicine C, Haemek Medical Center, Israel, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMC 70-16
Record Dates: First submitted 2016-10-27; First posted 2017-03-23 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hypomagnesemia
MeSH Terms: interventions — magnesium citrate; levulinic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): After initial intravenous treatment, participants (those with magnesium level ≥1 mg/dL) will be randomized, and oral magnesium therapy ( or no treatment) will be started. The experimental group will receive 400mg magnesium daily in two divided doses. Patients in the experimental group will be discharged with one month's supply of magnesium and continued for at least three months.
  Interventions: Drug: Magnesium Citrate 100 MG
- Control group (No Intervention): control group will receive standard care (no treatment). Patient will have their blood tested and will come for follow up visit every month for 3 months after discharge.

INTERVENTIONS:
Drug: Magnesium Citrate 100 MG — initial intravenous treatment: Patients with magnesium levels 1-1.5 mg/dL will receive 2-4 grams of magnesium sulfate in the first 24 hours. Patients with magnesium levels 1.6-1.9 mg/dL will receive 1 gram of magnesium sulfate. participants with magnesium level ≥1 mg/dL, will be randomized, and oral magnesium therapy, Magnesium Citrate, ( or no treatment) will be started, and continued for at least three months. The experimental group will receive 400mg magnesium daily in two divided doses.
  Other Names: Diasporal
  Arms: Experimental group

SUMMARY:
Hypomagnesemia is a common entity in the inpatient and outpatient setting. in previous retrospective study hypomagnesemic patients have higher mortality and longer hospitalization. whether hypomagnesemia is merely a marker of poor prognosis, or whether replacing it can improve outcomes is unclear. The current standard of care is to discharge these patients without workup or further treatment, even if patients had received intravenous therapy while hospitalized. The investigator wish to examine prospectively whether giving replacement therapy affects mortality, length of hospital stay and overall well-being. In order to replete intracellular levels and replete magnesium stores, magnesium should be given for several months.

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted over the age of 18, has hypomagnesemia (magnesium level ≤1.9 mg/dL) and is able to give consent.

Exclusion Criteria:

* A patient unable to give consent.
* A patient admitted for an elective procedure.
* A patient in critical condition or dying.
* Patients with advanced kidney disease with eGFR<15ml/min or on dialysis.
* Patients with severe diarrhea, precluding use of magnesium citrate.
* Patients already receiving magnesium supplements.
* Patients with severe malnutrition or life-threatening hypomagnesemia (serum level <1mg/dL), requiring intravenous and oral replacement of magnesium.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
compare mortality | one year
  To compare mortality between the population receiving magnesium and the population receiving standard care: ie no replacement.

SECONDARY OUTCOMES:
Hospitalization | one year
  Length in days of hospitalization.

OTHER OUTCOMES:
causes for hypomagnesemia | one year
  The investigators will attempt to ascertain the causes for hypomagnesemia from the data collected (medications, diarrhea, malnutrition, etc)
re-hospitalization | one year
  re-hospitalization for any cause
Subjective well-being | one year
  symptoms and overall well-being of the patients: a questionaire will be administered at the beginning of the study and at each visit regarding subjective feelings of well being, symptoms of pain, cramping and diarrhea, and overall functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Frieda Wolf, Principal Investigator — haemek medical center
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weglicki WB. Hypomagnesemia and inflammation: clinical and basic aspects. Annu Rev Nutr. 2012 Aug 21;32:55-71. doi: 10.1146/annurev-nutr-071811-150656. Epub 2012 Mar 8. PMID 22404119
- [Background] Rayssiguier Y, Libako P, Nowacki W, Rock E. Magnesium deficiency and metabolic syndrome: stress and inflammation may reflect calcium activation. Magnes Res. 2010 Jun;23(2):73-80. doi: 10.1684/mrh.2010.0208. Epub 2010 May 31. PMID 20513641
- [Background] Chaigne-Delalande B, Li FY, O'Connor GM, Lukacs MJ, Jiang P, Zheng L, Shatzer A, Biancalana M, Pittaluga S, Matthews HF, Jancel TJ, Bleesing JJ, Marsh RA, Kuijpers TW, Nichols KE, Lucas CL, Nagpal S, Mehmet H, Su HC, Cohen JI, Uzel G, Lenardo MJ. Mg2+ regulates cytotoxic functions of NK and CD8 T cells in chronic EBV infection through NKG2D. Science. 2013 Jul 12;341(6142):186-91. doi: 10.1126/science.1240094. PMID 23846901
- [Background] Misra PS, Alam A, Lipman ML, Nessim SJ. The relationship between proton pump inhibitor use and serum magnesium concentration among hemodialysis patients: a cross-sectional study. BMC Nephrol. 2015 Aug 13;16:136. doi: 10.1186/s12882-015-0139-9. PMID 26268579